CLINICAL TRIAL: NCT04925726
Title: Water-Based vs. Land-Based Rehabilitation After Arthroscopic Partial Meniscectomy in Middle-Aged Active Patients With a Degenerative Meniscal Tear: A Randomized, Controlled Study
Brief Title: Rehabilitation After Arthroscopic Partial Meniscectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hilal Yeşil (Other)
Responsible Party: Sponsor-Investigator, Hilal Yeşil, Assoc.Prof., Afyonkarahisar Health Sciences University
Organization: Afyonkarahisar Health Sciences University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MYHY
Record Dates: First submitted 2021-06-08; First posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Knee Pain
Keywords: Rehabilitation; Exercise; Aquatherapy
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Land based exercise (Active Comparator): Land based exercise
  Interventions: Other: Land based exercise
- Water based exercise (Active Comparator): Water based exercise
  Interventions: Other: Water based exercise

INTERVENTIONS:
Other: Land based exercise — The patients who had land based exercise
  Arms: Land based exercise
Other: Water based exercise — The patients who had water based exercise
  Arms: Water based exercise

SUMMARY:
Water-Based vs. Land-Based Rehabilitation After Arthroscopic Partial Meniscectomy in Middle-Aged Active Patients with a Degenerative Meniscal Tear: A Randomized, Controlled Study

DETAILED DESCRIPTION:
In this study, we aimed to determine and compare the benefits of water-based exercise (WBE) and land-based exercise (LBE) on pain, functionality, and quality of life after arthroscopic partial meniscectomy (APM). Middle-aged (35-50), active 30 patients having APM for a degenerative meniscal tear randomized into LBE (n=15) and WBE (n=15) groups. The pain level (visual analogue scale [VAS]), isokinetic muscle strength, quality of life (Short Form-36 [SF-36]), and function level (single-leg hop test and Lysholm questionnaire) were evaluated prior to treatment and at follow-up visits at the fourth and eighth week after surgery. The exercise sessions were conducted 3 times a week for 4 weeks in both groups.

ELIGIBILITY:
Inclusion Criteria: The inclusion criteria comprised a non-locked painful knee of more than 1 month, age between 35-50 years, a clinical history and examination compatible with degenerative meniscus, positive findings of a degenerative meniscal tear visible with magnetic resonance imaging (MRI), no response to nonoperative treatment of at least 3 months after onset of symptoms, and no evidence of advanced osteoarthritis (OA) on X-rays or MRI

Exclusion Criteria: The exclusion criteria employed were advanced knee OA, systemic inflammatory disease, a concurrent tear of posterior cruciate ligament, a concurrent collateral ligament repair, other problems causing knee pain (e.g., hip and ankle pathologies), a history of cardiopulmonary disease that could limit isokinetic and functional testing, an unstable medical condition, a serious cognitive deficit, a psychiatric problem, no capacity for independent walking and standing, an open wound on the skin, or pregnancy

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline VAS (visual analog scale) at 4th and 8th week | up to 8 weeks
  The patients were asked to make an assesment of their pain level between 0 and 10 scale

SECONDARY OUTCOMES:
Change from baseline isokinetic muscle strength at 4th and 8th week | up to 8 weeks
  Isokinetic knee extensor muscle strength of the patients was measured with an isokinetic dynamometer. The test was repeated 10 times at the velocity of 60°/second and 180°/second and peak torque (Nm) measurements were recorded .
Change from baseline quality of life (short form 36) at 4th and 8th week | up to 8 weeks
  The physical and mental health summary scores were the primary components used. Scoring is on a scale of 0 to 100 and a higher score reflects better health-related quality of life.
Change from baseline Single-leg hop test at 4th and 8th week | up to 8 weeks
  The patient stands on one foot with the big toe touching a line marked on the floor. The participant asked to hop forward as far as possible using the same leg with their arms swing freely on both sides of the body. Distance is measured from the starting point to the heel of the landing leg.
Change from baseline Lysholm questionnaire at 4th and 8th week | up to 8 weeks
  Eight subtitles are scored differently (limping or use of support: 5 points, locking sensation: 15 points, joint instability and pain: 25 points, swelling: 10 points, stair climbing: 10 points, and squatting: 5 points). The highest and optimal total score is 100 points

CONTACTS AND LOCATIONS:
Overall Officials: Murat Yesil, MD, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Hilal Yesil, Merkez, Afyonkarahisar, Turkey (Türkiye)

REFERENCES:
- [Derived] Yesil M, Ozcan O, Dundar U, Toktas H, Yesil H. Aquatic vs. land-based exercise after arthroscopic partial meniscectomy in middle-aged active patients with a degenerative meniscal tear: A randomized, controlled study. J Orthop Sci. 2023 Mar;28(2):391-397. doi: 10.1016/j.jos.2021.11.011. Epub 2021 Dec 16. PMID 34924251